CLINICAL TRIAL: NCT02494414
Title: Outcome of Cardiac Arrest Survivors: Prospective Cohort of Ile-de-France
Brief Title: Outcome of Cardiac Arrest Survivors
Acronym: DESAC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR12068
Record Dates: First submitted 2015-04-20; First posted 2015-07-10 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrest Survivors
Keywords: Cardiac arrest; outcome; neurological status
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- French prospective cohort of cardiac arrest survivors: Outcome of cardiac arrest survivors: prospective cohort of Ile-de-France
  Interventions: Other: Long-term follow-up

INTERVENTIONS:
Other: Long-term follow-up — Vital and neurological follow-up

SUMMARY:
Early prognosis of cardiac arrest - nearly 40000 new cases per year in France - has been extensively studied, highlighting a poor outcome (less than 8% at hospital discharge). However, little is known on mid and long-term prognostic factors and how these patients do survive from the event.

Using a regional cohort, the aim of the study is to describe long-term survival rate of cardiac arrest survivors, and to assess the influence of treatment strategies on survival and functional outcome.

DETAILED DESCRIPTION:
The collection of clinical and biological data of patients who experienced cardiac arrest and survive from hospital, including a regular follow-up with qualitative data (functional, neurological and quality of life) may provide important benchmark on the evolution of these patients and on the impact of acute interventions (such as cardio-pulmonary resuscitation, defibrillation, emergent coronary revascularization, neuroprotective treatments).

Using a large identified cohort of survivors of cardiac arrest, we aim to describe the qualitative long-term prognosis of these cardiac arrest patients (functional, neurological and quality of life status). Secondarily, we intend to identify the long-term prognostic factors, and particularly the role of early interventions, using a long-term and qualitative combined endpoint (vital status, functional scales, SF36).

This project is observational and will include all patients over 18 admitted alive after non-traumatic cardiac arrest in the area of Ile-de-France (France), whatever the cause of the cardiac arrest. Patients or their proxies, refusing their participation, will not be included.

We will collect all pre- and in-hospital information related to the event and performs prospectively interviews at 3 months and every year anniversary. The questionnaire will include vital status, cardiovascular events, medication and a complete qualitative report (SF36, ADL scale, OPC, CPC, social-professional activities).

This project will provide important data over time on the evolution of these patients. Findings will help in measuring the role of different strategies on long-term prognosis and consequently improve the overall management of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients alive after resuscitation from a out-of-hospital cardiac arrest
* All causes for cardiac arrest
* Age above 18
* Informed consent from the patient or next of kin

Exclusion Criteria:

* Impossibility for communication after hospital discharge, whatever the cause (language, residence…)
* Follow-up refusal from the patient or next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be prospectively included if they are discharged alive from intensive care after being resuscitated from a cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Cerebral Performance Categories Scale | at last follow-up (48 months max)
  Combined vital and neurological status

SECONDARY OUTCOMES:
SF-36 (Short-Form General Health Survey) | at last follow-up (48 months max)
  Quality of life
Overall Performance Categories (OPC) | at last follow-up (48 months max)
Activities of Daily Living (ADL) scale | at last follow-up (48 months max)
New cardiovascular events | at last follow-up (48 months max)
New York Heart Association (NYHA) status | at last follow-up (48 months max)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Empana, MD, Study Chair — INSERM U970 Centre de Recherche Cardiovasculaire de Paris Equipe 4, Epidémiologie Cardiovasculaire et Mort Subite
Locations (1):
- INSERM U970 Centre de Recherche Cardiovasculaire de Paris Equipe 4, Epidémiologie Cardiovasculaire et Mort Subite, Paris, France